CLINICAL TRIAL: NCT01441440
Title: A Randomized, Double-blind, Placebo Controlled, Multicenter Study To Evaluate The Efficacy And Safety Of Venlafaxine Er In Adult Outpatients With Major Depressive Disorder
Brief Title: Venlafaxine ER Phase 3 Study for Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2411263
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: venlafaxine ER; Major depressive disorder; Japan; placebo-controlled
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- venlafaxine ER 75 mg/day (fixed dose) (Experimental)
  Interventions: Drug: venlafaxine ER 75 mg/day (fixed dose)
- venlafaxine ER 75 mg/day to 225 mg/day (flexible dose) (Experimental)
  Interventions: Drug: venlafaxine ER 75 mg/day to 225 mg/day (flexible dose)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: venlafaxine ER 75 mg/day (fixed dose) — Treatment phase: 8 weeks (37.5 mg/day for 1st week and 75 mg/day for 7 weeks), oral administration Tapering phase: 2 weeks (37.5 mg/day for the 1st week and placebo for the 2nd week), oral administration
  Arms: venlafaxine ER 75 mg/day (fixed dose)
Drug: venlafaxine ER 75 mg/day to 225 mg/day (flexible dose) — Treatment phase: 8 weeks (37.5 mg/day for the 1st week, 75 mg/day for the 2nd weeks, 75-150 mg for the 3rd week, 75-225 mg/day for the rest of 5 weeks), oral administration Tapering phase: 2 weeks (75/37.5 mg/day for the 1st week and 37.5 mg/day/placebo for the 2nd week), oral administration
  Arms: venlafaxine ER 75 mg/day to 225 mg/day (flexible dose)
Drug: Placebo — Treatment phase: 8 weeks (placebo), oral administration Tapering phase: 2 weeks (placebo), oral administration
  Arms: Placebo

SUMMARY:
This is a phase 3, multi-center, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of venlafaxine ER 75 mg/day (fixed dose) and venlafaxine ER 75 mg/day to 225 mg/day (flexible dose), compared to placebo. This study consists of 2 week screening phase, 8 week treatment phase and 2 week tapering phase. The follow-up visit will be evaluated after 2 weeks of last study medication dosing.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient status.
* A primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM- IV-TR), single or recurrent episode, without psychotic features.
* Depressive symptoms for at least 90 days in single episode and for at least 28 days in recurrent episode before the screening visit.
* A MADRS total score ≥26 at the screening and baseline visits. And change of MADRS total score at baseline is not over 25% from the screening visit.
* A QIDS16-J-SR score ≥16 at the screening and baseline visits.
* A score ≥4 on the Clinical Global Impressions Scale-Severity (CGI-S) at the screening and baseline visits.

Exclusion Criteria:

* Subjects who concurrently have Axis II personality disorder or mental retardation according to DSM-IV diagnostic criteria.
* Subjects who meet DSM-IV criteria for current or past history of Schizophrenia, Paranoid Disorders, or any other Psychotic Disorders.
* Subjects who meet DSM-IV criteria for current or past history of Dementia.
* Subjects who meet DSM-IV criteria for current or past history of bipolar disorder, Posttraumatic Stress Disorder (PTSD) or Obsessive Compulsive Disorder (OCD).
* Subjects who meet DSM-IV criteria for current (within 12 months before the screening visit) generalized anxiety disorder, panic disorder, or social anxiety disorder considered by the investigator to be primary (causing a higher degree of distress or impairment than MDD).
* Subjects with a first degree relative with bipolar disorder.
* Subjects who are actively suicidal.
* History of non-responsive to 2 antidepressant treatment (at least 6-week usage for each) for the past or current episodes.
* History of Electroconvulsive therapy (ECT) at any time in the past.
* History of chronic treatment with benzodiazepines for longer than 6 months before the screening visit (Excluding subjects who have taken PRN benzodiazepine use, < 3 times/week).
* Any unstable hepatic, renal, pulmonary, cardiovascular (including uncontrolled hypertension), ophthalmologic, neurologic, or any other medical condition that in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of, the study.
* Known presence of raised intraocular pressure or history or presence of narrow angle glaucoma.
* Myocardial infarction within 180 days of the screening visit.
* Clinically important abnormalities, as determined by the investigator, on screening physical examination, electrocardiogram (ECG) or laboratory tests.
* Use of prohibited treatments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- Japan (63):
  - Narumi Himawari Clinic, Nagoya, Aichi-ken
  - Mizuho Clinic, Nagoya, Aichi-ken
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai, Chiba
  - Hida Clinic, Nagareyama, Chiba
  - Nakamoto Clinic, Noda, Chiba
  - Hatsuki Shinryo Clinic, Fukuoka, Fukuoka
  - Hatakeyama Clinic, Kitakyushu-shi, Fukuoka
  - Shiranui Hospital, Omuta, Fukuoka
  - Oka Clinic, Omuta, Fukuoka
  - Fujikawa Clinic, Hatsukaichi, Hiroshima
  - Hayakawa Clinic, Kure, Hiroshima
  - Kawamura Mental Clinic, Sapporo, Hokkaido
  - Maruyamapark Mentalclinic, Sapporo, Hokkaido
  - Arai Clinic, Amagasaki, Hyōgo
  - Takahashi Psychiatric Clinic, Ashiya, Hyōgo
  - Tatsuta Clinic, Kobe, Hyōgo
  - Ikeuchi Psycho Induced Internal Med.Clinic, Kobe, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Medical Corporation Seishinkai Kishiro Mental Clinic, Kawasaki, Kanagawa
  - Yutaka Clinic, Sagamihara, Kanagawa
  - Azamino Mental Clinic, Yokohama, Kanagawa
  - Shioiri Mental Clinic, Yokosuka, Kanagawa
  - Yuge Hospital, Kumamoto, Kumamoto
  - Kuginuki Clinic, Hirakata, Osaka
  - Shibamoto Clinic, Osakasayama-shi, Osaka
  - Sakai Mental Clinic, Saitama, Saitama
  - Suzuki Hospital, Adachi-ku, Tokyo
  - Iidabashi Mental Clinic, Chiyoda-ku, Tokyo
  - Tutujigaoka Mental Clinic, Chōfu, Tokyo
  - Fuku Clinic, Katsushika-ku, Tokyo
  - SAKURAZAKA CLINIC SophyAnce, Minato-ku, Tokyo
  - Akasaka Clinic, Minato-ku, Tokyo
  - Harikae mental clinic, Nakano-Ku, Tokyo
  - Heartcare Ginga Clinic, Nakano-ku, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Setagaya-ku, Tokyo
  - Komazawa Mental Clinic, Setagaya-ku, Tokyo
  - Omotesando Mental Clinic, Shibuya-ku, Tokyo
  - Maynds Tower Mental Clinic, Shibuya-ku, Tokyo
  - Yoyoginomori Mental Clinic, Shibuyaku, Tokyo
  - Meguro sta.East Mental Clinic, Shinagawa-ku, Tokyo
  - Himeno Tomomi Clinic, Shinagawa-Ku, Tokyo
  - Nishi-Shinjuku Concieria Clinic, Shinjuku-ku, Tokyo
  - Tamaki Clinic, Shinjuku-ku, Tokyo
  - Kagurazaka Stress Clinic, Shinjuku-ku, Tokyo
  - Tokyo Kosei Nenkin Hospital, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Himorogi Psychiatric Institute, Toshima-ku, Tokyo
  - Sugahara Tenjin Clinic, Fukuoka
  - Hiro Mental Clinic Tenjinminami, Fukuoka
  - Tenjin Mental Clinic, Fukuoka
  - Medical Corporation Shinseikai Kaku Mental Clinic, Fukuoka
  - Ange Psychiatric Clinic, Fukuoka
  - Stress Care Yoshimura Clinic, Fukuoka
  - Kuranari Psychiatry Clinic, Fukuoka
  - Akasaka Kato Clinic, Fukuoka
  - Imato Clinic, Fukuoka
  - Tsuji Mental Clinic, Hiroshima
  - Medical Corporation Toyokokai Tawara Clinic, Kanagawa
  - Sagaarashiyama-Tanaka Clinic, Kyoto
  - Kyo Mental Clinic, Nara
  - JIN clinic, Osaka
  - Misato Ekimae Clinic, Saitama
  - Eto Mental Clinic Meguro, Tokyo

REFERENCES:
- [Derived] Kato M, Asami Y, Wajsbrot DB, Wang X, Boucher M, Prieto R, Pappadopulos E. Clustering patients by depression symptoms to predict venlafaxine ER antidepressant efficacy: Individual patient data analysis. J Psychiatr Res. 2020 Oct;129:160-167. doi: 10.1016/j.jpsychires.2020.06.011. Epub 2020 Jul 9. PMID 32912597
- [Derived] Higuchi T, Kamijima K, Nakagome K, Itamura R, Asami Y, Kuribayashi K, Imaeda T. A randomized, double-blinded, placebo-controlled study to evaluate the efficacy and safety of venlafaxine extended release and a long-term extension study for patients with major depressive disorder in Japan. Int Clin Psychopharmacol. 2016 Jan;31(1):8-19. doi: 10.1097/YIC.0000000000000105. PMID 26513202
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2411263&StudyName=Venlafaxine%20ER%20Phase%203%20Study%20for%20Major%20Depressive%20Disorder%20%28MDD%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were confirmed to meet entry criteria at the screening visit, followed by a 2-week screening period. Subjects who continued to meet all study entry criteria at baseline were randomized to 10 weeks of treatment with placebo, venlafaxine ER 75 mg/day Fixed, or venlafaxine ER 75-225 mg/day Flexible in the ratio of 1:1:1.
Groups:
- Placebo: Participants received placebo capsule orally once daily after meal for 8 weeks.
- Venlafaxine 75 mg/Day Fixed: Participants received venlafaxine ER capsule orally once daily after meal for 8 weeks. Starting dose was 37.5 mg/day followed by 75 mg/day at Week 1. If there was no tolerability concern at Week 2, the dose was continued 75 mg/day until Week 8.
- Venlafaxine 75-225 mg/Day Flexible: Participants received venlafaxine ER capsule orally once daily after meal for 8 weeks. Starting dose was 37.5 mg/day followed by 75 mg/day at Week 1. If there was no tolerability concern at Week 2, the dose was increased to 150 mg/day. If there was no tolerability concern at Week 3, the dose was increased to 225 mg/day. Dose was reduced in the case of intolerability and if the participants could not take venlafaxine 75 mg/day or higher doses at Week 1 and the following weeks, the treatment were discontinued. No dose adjustment was allowed from Week 4 to Week 8.
Period: Overall Study
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Started | 183 (Safety analysis set) | 174 (Safety analysis set) | 180 (Safety analysis set)
Completed | 166 | 151 | 158
Not Completed | 17 | 23 | 22
Not completed — Death | 1 | 0 | 1
Not completed — Adverse Event | 2 | 9 | 9
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 11 | 9 | 9
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Moving | 0 | 1 | 1
Not completed — Work-related matter | 0 | 1 | 0
Not completed — Difficllty in keeping the schedule | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible | Total
Number analyzed (Participants) | 184 | 174 | 179 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.1) | 38.4 (11.9) | 38.3 (10.2) | 38.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 93 | 90 | 86 | 269
  MALE | 91 | 84 | 93 | 268

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 17-item Hamilton Raing Scale for Depression (HAM-D17) Total Score at Week 8 or Early Termination
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAM-D17 are rated on a scale of 0 to 2 or 0 to 4, and the total score ranges from 0 to 52. Higher scores indicate more severe symptoms. Change from baseline: mean score at Week 8 or early termination minus mean score at baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: Participants randomly assigned to treatment who took at least one dose of the study drug in the double-blind period and who had both baseline and at least one post-baseline measurements of the primary efficacy variable.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 184 | 174 | 177
Units on a scale | -9.25 (0.48) | -10.76 (0.50) | -10.37 (0.49)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.031, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [0.14 to 2.87] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.106, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-0.24 to 2.48] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

2. Secondary Outcome: Changes From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 8 or Early Termination
Description: MADRS is a scale used in subjects with major depressive disorder to measure the overall severity of depressive symptoms. It is a 10 item, clinician-rated scale that assesses treatment-sensitive change by evaluating ten areas of depressive symptomatology: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts. The items are rated on a 7 point Likert scale (0 - 6) with anchors at 2 point intervals. The total score ranges from 0 to 60, and higher scores indicate more severe symptoms. Change from baseline: mean score at Week 8 or early termination minus mean score at baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 182 | 172 | 176
Units on a scale | -12.41 (0.75) | -15.30 (0.77) | -15.05 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.008, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 2.88, 95% CI 2-sided [0.77 to 5.00] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.014, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 2.64, 95% CI 2-sided [0.54 to 4.74] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

3. Secondary Outcome: Changes From Baseline in Clinical Global Impression-Severity (CGI-S) at Week 8 or Early Termination
Description: CGI-S is a 7-point clinician rated scale to assess severity of participant's current illness state; range: 1=normal, not ill at all, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill patients. Higher scores reflect higher severity of current illness states. Change from baseline: mean score at Week 8 or early termination minus mean score at baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 184 | 174 | 177
Units on a scale | -1.31 (0.08) | -1.57 (0.08) | -1.56 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.025, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.03 to 0.49] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.032, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.02 to 0.48] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

4. Secondary Outcome: Changes From Baseline in 6-item Hamilton Rating Scale for Depression (HAM-D6) Total Score at Week 8 or Early Termination
Description: HAM-D6 is a subset of the HAM-D17 that assesses 6 items associated with major depression. The scale uses HAM-D17 items 1, 2, 7, 8, 10 and 13. Item 13 is scored 0 to 2 and all others are scored 0 to 4. Total score ranges from 0 to 22; higher score indicates more depression. Change from baseline: mean score at Week 8 or early termination minus mean score at baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 184 | 174 | 177
Units on a scale | -4.92 (0.28) | -6.10 (0.29) | -5.99 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.004, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [0.39 to 1.97] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.008, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [0.28 to 1.85] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

5. Secondary Outcome: Changes From Baseline in 16-item Quick Inventory of Depressive Symptomatology Self-Report Japanese Version (QIDS16-SR-J) Total Score at Week 8 or Early Termination
Description: QIDS16-SR-J is a self-rated scale used in patients with major depressive disorder to measure the overall severity of depressive symptoms: 1) sad mood; 2) concentration; 3) self-criticism; 4) suicidal ideation; 5) interest; 6) energy/fatigue; 7) sleep disturbance (initial, middle, and late insomnia or hypersomnia); 8) decrease/increase in appetite/weight; and 9) psychomotor agitation/retardation. QIDS16-SR-J items are rated on a scale of 0 to 3. The total score ranges from 0 to 27, and higher scores indicate more severe symptoms. Change from baseline: mean score at Week 8 or early termination minus mean score at baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 182 | 172 | 175
Units on a scale | -6.50 (0.36) | -8.00 (0.37) | -7.27 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.004, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [0.48 to 2.53] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.137, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline as a covariate; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.25 to 1.79] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

6. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Score at Week 8 or Early Termination
Description: CGI-I is a 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Scores above 4 reflect worsening of illness state as compared to baseline.
Time Frame: Baseline, Week 8 or Early termination
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Number analyzed (Participants) | 184 | 174 | 177
Units on a scale | 2.53 (0.08) | 2.32 (0.09) | 2.28 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Venlafaxine 75 mg/Day Fixed; Test type: Superiority or Other; p = 0.073, ANCOVA — Two-sided p-value from an analysis of covariance model including treatment as a factor and baseline score of CGI-S as a covariate; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.02 to 0.45] — Adjusted mean difference = Placebo group - Venlafaxine 75 mg/day Fixed group
Statistical Analysis 2: Comparison: Placebo vs Venlafaxine 75-225 mg/Day Flexible; Test type: Superiority or Other; p = 0.034, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.02 to 0.48] — Adjusted mean difference = Placebo group - Venlafaxine 75-225 mg/day Flexible group

ADVERSE EVENTS:
Arm/Group | Placebo | Venlafaxine 75 mg/Day Fixed | Venlafaxine 75-225 mg/Day Flexible
Serious Adverse Events (participants affected / at risk) | 2/183 | 1/174 | 1/180
Other Adverse Events (participants affected / at risk) | 98/183 | 112/174 | 131/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=183) | Venlafaxine 75 mg/Day Fixed (N=174) | Venlafaxine 75-225 mg/Day Flexible (N=180)
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=183) | Venlafaxine 75 mg/Day Fixed (N=174) | Venlafaxine 75-225 mg/Day Flexible (N=180)
Palpitations (Cardiac disorders) | 5 | 8 | 6
Tachycardia (Cardiac disorders) | 0 | 4 | 7
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 6
Abdominal discomfort (Gastrointestinal disorders) | 4 | 7 | 11
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5 | 0
Constipation (Gastrointestinal disorders) | 8 | 17 | 17
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 5 | 7
Nausea (Gastrointestinal disorders) | 24 | 39 | 53
Vomiting (Gastrointestinal disorders) | 7 | 5 | 4
Feeling abnormal (General disorders) | 0 | 2 | 4
Malaise (General disorders) | 5 | 9 | 11
Thirst (General disorders) | 14 | 11 | 18
Nasopharyngitis (Infections and infestations) | 41 | 35 | 32
Alanine aminotransferase increased (Investigations) | 0 | 4 | 2
Blood pressure increased (Investigations) | 2 | 4 | 5
Heart rate increased (Investigations) | 4 | 10 | 13
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 4
Dizziness (Nervous system disorders) | 5 | 10 | 18
Dizziness postural (Nervous system disorders) | 1 | 2 | 5
Headache (Nervous system disorders) | 14 | 16 | 18
Somnolence (Nervous system disorders) | 15 | 21 | 31
Insomnia (Psychiatric disorders) | 6 | 4 | 8
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.